CLINICAL TRIAL: NCT01276886
Title: Italian Study Group on Complicated Diverticulosis: The Natural History of Left-sided Acute Diverticulitis
Brief Title: Italian Study Group on Complicated Diverticulosis
Acronym: GISDIC
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano per lo Studio della Diverticolite Complicata (Other)
Other Study IDs: GISDIC-1
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-12

CONDITIONS: Diverticulitis
Keywords: Left sided acute diverticulitis diagnosed clinically by the presence of abdominal pain, leukocytosis (>11x109) and/or fever >38°C, confirmed by imaging.; CT criteria: localized thickening (≥4 mm) of the colonic wall and signs of inflammation of the pericolic fat, abscess and/or extraluminal air and/or contrast.; US criteria: bowel wall thickening (>4 mm), diverticular inflammation, pericolic fat edema, intramural or pericolic inflammatory mass, intramural fistula.; WSCE criteria: segmental luminal narrowing and a tethered mucosa with or without a mass effect or extravasation of contrast and/or extraluminal air.
MeSH Terms: conditions — Diverticulitis; Leukocytosis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Diverticulitis
  Interventions: Drug: antibiotic; Procedure: Colonic resection with or without stoma

INTERVENTIONS:
Drug: antibiotic
Procedure: Colonic resection with or without stoma

SUMMARY:
Patients were recruited over a four year period from 1996 to 1999. Those admitted in the years 1996 and 1997 were retrospectively accrued from the clinical records, while patients treated between 1998 and 1999 patients were entered on the database prospectively on admission.

Inclusion criteria All consecutive patients with left sided acute diverticulitis diagnosed clinically by the presence of abdominal pain, associated with leukocytosis (>11x109) and/or fever >38°C, confirmed by imaging (CT scan, ultrasonography, water soluble contrast enema) either alone or in combination and/or by operative findings, entered the study. The CT criteria for the diagnosis included a localized thickening (≥4 mm) of the colonic wall and signs of inflammation of the pericolic fat, with abscess and/or extraluminal air and/or extraluminal contrast. The criteria for ultrasound included at least two of the following signs: bowel wall thickening (>4 mm), diverticular inflammation, pericolic fat edema, intramural or pericolic inflammatory mass, intramural fistula. The diagnostic criteria for water soluble contrast enema included segmental luminal narrowing and a tethered mucosa with or without a mass effect or extravasation of contrast and/or the presence of extraluminal air.

Exclusion criteria Patients with inflammatory bowel disease, irritable bowel syndrome, colorectal cancer or diseases precluding adequate follow up, were excluded from the study.

Treatment Patients were treated conservatively (antibiotics, I.V. nutrition, CT/US guided abscess drainage) or surgically according to the local policy of each center.

Follow up Follow up was carried out according to local policy. The following data were collected: persistence or recurrence of chronic symptoms attributable to complicated diverticular disease, new episodes of AD, new hospital admissions for AD, type of treatment and outcome.

Recurrence was defined as a new episode of AD requiring hospitalization that occurred at least 2 months after complete resolution of the index episode which resulted in inclusion in the study. If surgery was performed, the timing, type of procedure, Hinchey stage and complications were recorded.

Data collection A standardized flow sheet was used to collect data on medical history, diagnostic work up, type of treatment and follow up to create a dedicated database. Gender, age, date of hospital admission and discharge, diagnosis on admission and discharge, co-morbidities (diabetes mellitus, cardiovascular disease, atherosclerosis, liver or renal failure), symptoms experienced before admission and their duration, history of diverticulosis, previous episodes of AD, laboratory tests, and treatment performed were recorded. Where surgery was performed, the date and type of procedure, the operative findings including Hinchey's classification (16) and details of the operation (incision, extension of resection, type of anastomosis, covering stoma, drains), pathology report, and postoperative complications occurring within 30 days, were all recorded.

End points The primary endpoint was to assess the rate of recurrence of AD requiring hospitalization during the follow-up period. Additional endpoints were to assess the risks of emergency surgery, stoma and disease-related mortality during the follow up.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with left sided acute diverticulitis diagnosed clinically by the presence of:

* abdominal pain,
* leukocytosis (>11x109)
* fever >38°C and confirmed by imaging (CT scan, ultrasonography, water soluble contrast enema)

The CT criteria for the diagnosis included at least one of:

* a localized thickening (≥4 mm) of the colonic wall
* signs of inflammation of the pericolic fat
* abscess
* extraluminal air
* extraluminal contrast

The ultrasound criteria included at least two of:

* bowel wall thickening (>4 mm)
* diverticular inflammation
* pericolic fat edema
* intramural or pericolic inflammatory mass
* intramural fistula

Water soluble contrast enema criteria included at least two of:

* segmental luminal narrowing
* a tethered mucosa
* a mass effect
* extravasation of contrast
* the presence of extraluminal air

Exclusion Criteria:

* inflammatory bowel disease
* irritable bowel syndrome
* colorectal cancer
* diseases precluding adequate follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients with left sided acute diverticulitis diagnosed clinically by the presence of abdominal pain, associated with leukocytosis (>11x109) and/or fever >38°C, confirmed by imaging (CT scan, ultrasonography, water soluble contrast enema) either alone or in combination and/or by operative findings
Sampling Method: Non-Probability Sample
Dates: Start 1996-01; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
to assess the rate of recurrence of acute diverticulitis requiring hospitalization during the follow-up period | 10 years

SECONDARY OUTCOMES:
to assess the risks of emergency surgery, stoma and disease-related mortality during the follow up | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery - Galliera Hospital, Genova, Italy